CLINICAL TRIAL: NCT05662202
Title: A Randomized, Double-blind, Vehicle-controlled, Multicenter Phase III Study to Evaluate the Safety, Tolerability, and Efficacy of BF-200 ALA (Ameluz®) in the Field-directed Treatment of Actinic Keratosis on the Extremities and Neck/Trunk With Photodynamic Therapy (PDT) Using the BF-RhodoLED® XL or BF-RhodoLED® Lamp
Brief Title: Study to Evaluate the Safety, Tolerability and Efficacy of BF-200 ALA (Ameluz®) in the Field-directed Treatment of Actinic Keratosis (AK) on the Extremities and Neck/Trunk With Photodynamic Therapy (PDT) Using a RhodoLED Lamp
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biofrontera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALA-AK-CT019
Record Dates: First submitted 2022-11-29; First posted 2022-12-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Actinic Keratoses
Keywords: Actinic keratosis; Photodynamic therapy; 5-aminolevulinic acid; Photosensitizing Agents
MeSH Terms: conditions — Keratosis, Actinic | interventions — BF-200 ALA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- BF-200 ALA (Experimental): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  Red light photodynamic therapy (PDT)
  Interventions: Combination Product: BF-200 ALA and red light LED lamp
- Vehicle (Placebo Comparator): Topical application of vehicle to BF-200 ALA containing no active ingredient. Red light photodynamic therapy (PDT)
  Interventions: Combination Product: Vehicle and red light LED lamp

INTERVENTIONS:
Combination Product: BF-200 ALA and red light LED lamp — Up to two PDTs using a RhodoLED lamp (RhodoLED® XL or BF-RhodoLED®) (ALA-PDT, Ameluz®-PDT):
  Topical application of up to 3 tubes BF-200 ALA on the expanded treatment field (up to 240 cm²), followed by red light illumination with a RhodoLED lamp after 3 h incubation of study medication under occlusive dressing.
  PDT-1 will be performed at Visit 2. Clinical clearance will be assessed 12 weeks after PDT-1 (Visit 4). In case of remaining lesions at Visit 4, PDT-2 will be performed at the same visit.
  Arms: BF-200 ALA
Combination Product: Vehicle and red light LED lamp — Up to two PDTs using a RhodoLED lamp (RhodoLED® XL or BF-RhodoLED®) (Vehicle-PDT):
  Topical application of up to 3 tubes vehicle on the expanded treatment field (up to 240 cm²), followed by red light illumination with a RhodoLED lamp after 3 h incubation of study medication under occlusive dressing.
  PDT-1 will be performed at Visit 2. Clinical clearance will be assessed 12 weeks after PDT-1 (Visit 4). In case of remaining lesions at Visit 4, PDT-2 will be performed at the same visit.
  Arms: Vehicle

SUMMARY:
The aim of this study is to test the safety. tolerability and efficacy of field-directed photodynamic therapy (PDT) with 10% aminolevulinic acid gel (Ameluz®, BF-200 ALA) in combination with one of the narrow spectrum red light RhodoLED lamps in comparison to vehicle treatment for actinic keratosis (AK) on the extremities and neck/trunk.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability of subjects to provide informed consent and sign the Health Insurance Portability and Accountability Act (HIPAA) form. A study-specific informed consent and HIPAA form must be obtained in writing prior to starting any study procedures.
2. 4 - 15 mild to moderate clinically confirmed AK lesions according to Olsen either on the extremities or on the neck/trunk with a diameter of ≥ 4 mm that must be present in the treatment field (defined as AK target lesions). In addition, non-target AK lesions may be present in the treatment field, including up to two severe AK lesions ≥ 4 mm. For each severe AK lesion (≥ 4 mm), a biopsy must be taken for confirmation of diagnosis. The treatment field (continuous or in several patches) totaling approx. either 80 cm², 160 cm² or 240 cm2 must be within one effective illumination area of the BF-RhodoLED® XL but may require up to three illuminations with the BF-RhodoLED®. All AK target lesions and, if applicable, severe AK lesions ≥ 4 mm located in the treatment field should be clearly distinguishable, without restrictions on the distance between lesions, and should have a minimal distance of 1 cm to the border of the treatment field.
3. All sexes, ≥ 18 years of age.
4. Willingness to undergo a 2 mm punch biopsy for each (up to two) severe AK lesion ≥ 4 mm, if applicable, at the screening visit.
5. Willingness and ability to comply with study procedures, particularly willingness to receive up to 2 PDTs within approximately 12 weeks.
6. Subjects with good general health or with clinically stable medical conditions will be permitted to be included in the study.
7. Willingness to stop the use of moisturizers and any other non-medical topical treatments within the treatment field at least 24 h prior to the next clinical visit.
8. Acceptance to abstain from extensive sunbathing and the use of a solarium or tanning beds during the treatment phase.
9. For female subjects with reproductive potential: Negative serum pregnancy test.
10. For female subjects with reproductive potential: Effective contraception at screening visit and throughout the treatment phase of the study (until Visit 4 or Visit 6).

Exclusion Criteria:

1. Any known history of hypersensitivity to ALA, porphyrins, or excipients of BF-200 ALA.
2. History of soy or peanut allergy.
3. Sunburn or other possible confounding skin conditions (e.g., wounds, irritations, bleeding, or skin infections) inside or in close proximity (< 2 cm distance) to the treatment field.
4. Clinically significant (cs) medical conditions making implementation of the protocol or interpretation of the study results difficult or impairing subject's safety such as:

   1. Presence of photodermatoses or porphyria
   2. Metastatic tumor or tumor with high probability of metastasis
   3. Infiltrating skin neoplasia (suspected or known)
   4. Unstable cardiovascular disease (New York Heart Association class III, IV)
   5. Unstable hematologic (including myelodysplastic syndrome), hepatic, renal, neurologic, or endocrine condition
   6. Unstable collagen-vascular condition
   7. Unstable gastrointestinal condition
   8. Immunosuppressive condition
   9. Presence of clinically significant inherited or acquired coagulation defect
5. Clinical diagnosis of atopic dermatitis, Bowen´s disease (BD), basal cell carcinoma (BCC), eczema, psoriasis, rosacea, squamous cell carcinoma (SCC), other malignant or benign tumors inside or in close proximity (< 2 cm distance) to the treatment field.
6. Presence of strong artificial pigmentation (e.g., tattoos) or any other abnormality that may impact lesion assessment or light penetration in the treatment field.
7. Any physical therapy such as cryotherapy, laser therapy, electrodessication, microdermabrasion, surgical removal of lesions, curettage, or treatment with chemical peels such as trichloroacetic acid inside or in close proximity (< 10 cm distance) to the treatment field within 4 weeks prior to screening.
8. Any of the topical treatments defined below within the designated periods prior to screening:

   1. Topical treatment with ALA or ALA esters (e.g., methyl aminolevulinic acid (MAL)) inside the treatment field within 3 months.
   2. Topical treatment with immunomodulatory, cytostatic, or cytotoxic drugs inside or in close proximity (< 10 cm distance) to the treatment field within 3 months.
   3. Start of topical administration of a medication with hypericin or other drugs with phototoxic or photoallergic potential inside or in close proximity (< 10 cm distance) to the treatment field within 4 weeks. Subjects may, however, be eligible if such medication was applied for more than 4 weeks prior to screening without evidence of an actual phototoxic/photoallergic reaction.
9. Any use of the systemic treatments within the designated periods prior to screening:

   1. Cytostatic or cytotoxic drugs within 6 months.
   2. Immunosuppressive therapies or ALA or ALA esters (e.g., MAL) within 12 weeks.
   3. Drugs known to have major organ toxicity within 8 weeks.
   4. Interferon or glucocorticosteroids within 6 weeks.
   5. Start of intake of medication with hypericin or drugs with phototoxic or photoallergic potential within 8 weeks prior to screening. Subjects may, however, be eligible if such medication was taken in for more than 8 weeks prior to the screening visit without evidence of an actual phototoxic/photoallergic reaction.
10. Breast feeding women.
11. Suspicion of drug or alcohol abuse.
12. Subjects unlikely to comply with protocol, e.g., inability to return for visits, unlikely to complete the study, or inappropriate in the opinion of the investigator.
13. A member of study site staff or sponsor staff directly involved in the conduct of the protocol or a close relative thereof.
14. Receipt of any investigational drug or medical product within 8 weeks before screening or simultaneous participation in another clinical study.

Reassessment of subjects is allowed once in case exclusion criterion 3 is met and eligibility can be achieved within 4 weeks. Reassessment can be done on the day of the actual treatment.

Dosing day exclusion criteria:

At Visit 2 (baseline, PDT-1)

Subjects with sunburn or other possibly confounding skin conditions (e.g., wounds, irritations, bleeding, or skin infections) inside or in close proximity (< 2 cm distance) to the treatment field. Reassessment of subjects is allowed once if the sunburn or other confounding skin conditions is/are expected to resolve within 2 weeks.

At Visit 4 (PDT-2)

Subjects with sunburn or other possibly confounding skin conditions (e.g., wounds, irritations, bleeding, or skin infections) inside or in close proximity (< 2 cm distance) to the treatment field. Rescheduling of PDT-2 can be performed once at the earliest possibility after resolution, but rescheduling should not exceed 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall subject complete response rate | 12 weeks after the last PDT (Visit 4 or Visit 6)
  Percentage of subjects with all AK target lesions clinically cleared after last PDT

SECONDARY OUTCOMES:
Overall subject complete response rate for subjects with lesions treated on extremities | 12 weeks after the last PDT (Visit 4 or Visit 6)
  Percentage of subjects with all AK target lesions on extremities clinically cleared after last PDT
Overall subject complete response rate for subjects with lesions treated on neck/trunk | 12 weeks after the last PDT (Visit 4 or Visit 6)
  Percentage of subjects with all AK target lesions on neck/trunk clinically cleared after last PDT
Lesion complete response rate | 12 weeks after the last PDT (Visit 4 or Visit 6)
  Percentage of clinically cleared individual AK target lesions in relation to total number of AK target lesions at baseline (Visit 2) after the last PDT, overall and stratified by treatment area and AK severity at baseline (according to Olsen)
Complete response rate for severe lesions | 12 weeks after the last PDT (Visit 4 or Visit 6)
  Percentage of clinically cleared individual severe AK lesions in relation to total number of severe AK lesions at baseline (according to Olsen; Visit 2) after the last PDT, overall and stratified by treatment area
Subject complete response rate after PDT-1 | 12 weeks after PDT-1 (Visit 4)
  Percentage of subjects with all AK target lesions clinically cleared after PDT-1, overall and stratified by AK baseline parameters
Lesion complete response rate after PDT-1 | 12 weeks after PDT-1 (Visit 4)
  Percentage of clinically cleared individual AK target lesions in relation to total number of AK target lesions at baseline (Visit 2) after PDT-1, overall and stratified by treatment area and AK severity at baseline (according to Olsen [mild, moderate, severe])
Complete response rate for severe lesions after PDT-1 | 12 weeks after PDT-1 (Visit 4)
  Percentage of clinically cleared individual severe AK lesions in relation to total number of severe AK lesions at baseline (according to Olsen [mild, moderate, severe]; Visit 2) after PDT-1, overall and stratified by treatment area
Esthetic appearance at the end of treatment phase assessed by the investigator | On final visit of the treatment phase, 12 weeks after the last PDT (Visit 4 or Visit 6)
  The esthetic appearance after the last PDT as assessed by the investigator as assessed by the subject according to a 4-point scale ranging from 0 (=very good) to 3 (=unsatisfactory); overall and stratified by treatment area
Esthetic outcome at the end of treatment phase assessed by the subject | On final visit of the treatment phase, 12 weeks after the last PDT (Visit 4 or Visit 6)
  The esthetic outcome after the last PDT as assessed by the subject according to a 4-point scale ranging from 0 (=very good) to 3 (=unsatisfactory); overall and stratified by treatment area
Satisfaction with PDT at the end of treatment phase | On final visit of the treatment phase, 12 weeks after the last PDT (Visit 4 or Visit 6)
  Satisfaction with PDT treatment after the last PDT as assessed by the subject via questionnaire, 1. if they would chose PDT treatment in the future in case of recurrence or similar disease (yes/no) and 2. how they would rate the PDT treatment in comparison to other treatment modalities, if applicable (better than/ similar/ worse). The treatment modalities should be documented, if applicable); overall and stratified by treatment area
Frequency and extent of adverse events (AEs), AEs of Special Interest (AESIs), serious AEs (SAEs) and treatment-emergent AEs (TEAEs) during treatment phase | Entire study duration, approx. 16 weeks for subjects requiring 1 PDT (until Visit 4) and approx. 28 weeks for subjects with 2 PDTs (until Visit 6)
  Frequency and extent of AEs, AESIs, SAEs, and TEAEs, overall and stratified by demographics, skin type class (I-III and IV-VI), size of the treatment field, and treatment area.
  TEAEs (including application site skin reactions and discomfort) are defined as all AEs with onset or worsening after treatment with IMP.
New lesions inside the treatment field during treatment phase | All clinical visits throughout entire study duration, approx. 16 weeks for subjects requiring 1 PDT (until Visit 4) and approx. 28 weeks for subjects with 2 PDTs (until Visit 6)
  New lesions: AK, non-melanoma skin cancer [NMSC, including Basal Cell Carcinoma (BCC), Squamous Cell Carcinoma (SCC) or Bowen's Disease (BD)] or melanoma
Assessment of application site reactions | All visits (except screening, Visit 1) throughout entire study duration, approx. 16 weeks for subjects requiring 1 PDT (until Visit 4) and approx. 28 weeks for subjects with 2 PDTs (until Visit 6)
  Application site reactions (bleeding, burning, discharge, edema, erosion, erythema, exfoliation, hyperalgesia, induration, irritation, paraesthesia, pruritus, pustules, scabbing, or vesicles) will be assessed on a 4-point scale: grade 0 = none, grade 1 = mild, grade 2 = moderate, grade 3 = severe.
Application site pain during illumination | During treatment (illumination) on treatment day for PDT-1 (Visit 2, up to 4 weeks after screening) and during treatment (illumination) on treatment day for PDT-2 (Visit 4; if applicable; 12 weeks after PDT-1)
  Reported by the subjects assessed on an 11-point numeric rating scale ranging from 0 (no pain) to 10 (worst imaginable pain); overall and stratified by size of the treatment field and treatment area
Number of patients with significant changes of vital signs | All clinical visits throughout entire study duration, approx. 16 weeks for subjects requiring 1 PDT (until Visit 4) and approx. 28 weeks for subjects with 2 PDTs (until Visit 6)
  Number of patients with changes in blood pressure (systolic and diastolic) [mmHg] and changes in pulse rate [beats/min]. Findings which differ from reference range and are considered to be clinically significant are to be reported.
Number of patients with significant changes in safety laboratory | All clinical visits throughout entire study duration, approx. 16 weeks for subjects requiring 1 PDT (until Visit 4) and approx. 28 weeks for subjects with 2 PDTs (until Visit 6)
  Changes in clinical chemistry, in hematology and urinalysis parameters as defined in the protocol. Findings which differ from reference range and are considered to be clinically significant are to be reported.
Number of patients with abnormal findings in physical examination | At screening (up to 4 weeks before treatment) and 12 weeks after the last PDT (Visit 4 or Visit 6)
  Physical examination of head, neck, skin, lymph nodes, thorax including heart and lungs, abdomen, and musculoskeletal, peripheral vascular and nervous system status will be performed. Abnormal findings, considered to be clinically significant, are to be reported.

OTHER OUTCOMES:
Subject recurrence rate | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  The percentage of subjects with all AK target lesions clinically cleared 12 weeks after the last PDT presenting with at least one recurrent lesion during follow-up, stratified by demographics, study sites, AK baseline parameters
Lesion recurrence rate | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  The percentage of AK target lesions showing recurrence in follow-up in relation to total number of clinically cleared AK target lesions 12 weeks after last PDT; overall and stratified by treatment area and AK severity at baseline (according to Olsen [mild, moderate, severe])
Recurrence rate of severe lesions | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  The percentage of severe AK lesions (according to Olsen [mild, moderate, severe]) showing recurrence in follow-up in relation to total number of clinically cleared severe AK lesions 12 weeks after last PDT; overall and stratified by treatment area
Esthetic appearance at follow-up visits assessed by the investigator | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  The esthetic outcome at follow-up visits as assessed by the subject according to a 4-point scale ranging from 0 (=very good) to 3 (=unsatisfactory); overall and stratified by treatment area
Esthetic outcome at follow-up visits assessed by the subject | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  The esthetic outcome at follow-up visits as assessed by the subject according to a 4-point scale ranging from 0 (=very good) to 3 (=unsatisfactory); overall and stratified by treatment area
Satisfaction with PDT at follow-up visits | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  Satisfaction with PDT treatment after the last PDT as assessed by the subject via questionnaire, 1. if they would chose PDT treatment in the future in case of recurrence or similar disease (yes/no) and 2. how they would rate the PDT treatment in comparison to other treatment modalities, if applicable (better than/ similar/ worse). The treatment modalities should be documented, if applicable); overall and stratified by treatment area
Any SAE and relevant AE | Entire follow-up duration, approx. 40 weeks
  Relevant AEs include AEs or conditions affecting skin health in the treatment field which may impair proper assessment of the recurrence rate of the treated AK lesions, or other clinically relevant events at the investigator's discretion as well as any SAE that has occurred since the final visit of the treatment phase (Visit 4 or Visit 6); overall and stratified by demographics and treatment area
New lesions inside the treatment field during follow-up | On follow-up Visit 1 (6 months after last PDT) and follow-up Visit 2 (12 months after last PDT)
  New lesions: AK, non-melanoma skin cancer [NMSC, including BCC, SCC or BD] or melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Zeitouni, MD, Principal Investigator — Medical Dermatology Specialists; Phoenix, Arizona, United States
Locations (14):
- United States (14):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Alliance Dermatology & Mohs Center, Phoenix, Arizona
  - Dermatology Practice, Greenwood Village, Colorado
  - Dermatology Associates PA of the Palm Beaches, Delray Beach, Florida
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Laser and Skin Surgery Center of Indiana, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Skin Search of Rochester, Inc., Rochester, New York
  - Rochester Dermatologic Surgery, Victor, New York
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - DermResearch, P.A., Austin, Texas
  - Austin Institute for Clinical Research, Houston, Texas
  - Austin Institute for Clinical Research Inc., Pflugerville, Texas